CLINICAL TRIAL: NCT00377403
Title: Randomized Clinical Trial to Evaluate Guidelines for Acute Rhinosinusitis (Phase IV Study)
Brief Title: Treatment of Acute Sinusitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Jane Garbutt, MD, Associate Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-0140; U01AI064655-01A1 (NIH)
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Results first posted 2011-06-29 (Estimated); Last update posted 2012-12-28 (Estimated); Status verified 2012-12

CONDITIONS: Acute Respiratory Infections; Acute Rhinosinusitis
Keywords: rhinosinusitis, sinusitis, amoxicillin
MeSH Terms: conditions — Rhinosinusitis; Sinusitis | interventions — Acetaminophen; Amoxicillin; Dextromethorphan; Guaifenesin; Acetylcysteine; Pseudoephedrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Arm (Experimental): Amoxicillin 500mg three times a day (tid) for 10 days in addition to symptomatic treatments
  Interventions: Drug: Acetaminophen; Drug: Amoxicillin; Drug: Dextromethorphan hydrobromide with guaifenesin; Drug: Guaifenesin; Drug: Pseudoephedrine Sustained Action; Drug: Saline spray (0.65%)
- Symptomatic treatments only (Placebo Comparator): Placebo for 10 days in addition to symptomatic treatments
  Interventions: Drug: Acetaminophen; Drug: Dextromethorphan hydrobromide with guaifenesin; Drug: Guaifenesin; Drug: Pseudoephedrine Sustained Action; Drug: Saline spray (0.65%)

INTERVENTIONS:
Drug: Acetaminophen — Symptomatic treatment:
  Dose: 500mg every 4 to 6 hours for pain or fever
  Other Names: Tylenol
Drug: Amoxicillin — Intervention drug:
  Dose: 500mg tid for 10 days
  Other Names: Amoxil
  Arms: Intervention Arm
Drug: Dextromethorphan hydrobromide with guaifenesin — Symptomatic treatment:
  Dose: 10mls every 4 to 6 hours for cough
  Other Names: Robitussin
Drug: Guaifenesin — Symptomatic treatment:
  Dose: 600mg every 12 hours to thin secretions
  Other Names: Mucinex OTC
Drug: Pseudoephedrine Sustained Action — Symptomatic treatment:
  Dose: 120mg every 12 hours for nasal congestion
  Other Names: Sudafed
Drug: Saline spray (0.65%) — Symptomatic treatment:
  Dose: 2 squeezes per nostril as needed for nasal congestion
  Other Names: Ocean Nasal Spray

SUMMARY:
This study will compare the symptom relief provided by 5 cold medicines versus the symptom relief provided by the same 5 cold medicines plus the antibiotic, amoxicillin, in people who have sinus infections. Treatment with amoxicillin may be more effective than treatment with cold medicines alone. Two hundred adult volunteers, aged 18 to 70 years old, with sinus infections will participate in this study for 28 days. Volunteers will receive a 10-day course of either amoxicillin or placebo (substance containing no medication). In addition, all volunteers will receive pain medication, a chest decongestant, nasal decongestants, and cough medicine as needed. Volunteers will be interviewed by telephone on days 0, 3, 7, 10, and 28 following the start of treatment. The study will look at quality of life factors such as change in functional status (ability to perform daily activities) and symptoms, recurrence of the infection, satisfaction with care, and the direct costs of treatment.

DETAILED DESCRIPTION:
The primary objective of this phase IV, randomized, placebo controlled clinical trial is to determine the incremental effect of amoxicillin treatment compared with symptomatic treatments on disease-related quality of life in adults with clinically diagnosed acute bacterial rhinosinusitis. The secondary objective is to determine the incremental effect of amoxicillin treatment compared with symptomatic treatments on functional status, symptoms, disease recurrence, satisfaction with treatment, and direct costs of treatment in adults with clinically diagnosed acute bacterial rhinosinusitis. The tertiary objective is to identify prognostic indicators for clinical improvement with antibiotic treatment in adults with clinically diagnosed acute bacterial rhinosinusitis. Two hundred adult subjects, 18 to 70 years old, who meet the recommended criteria for acute bacterial rhinosinusitis, will be enrolled from 8 practice sites. Subjects will be randomized to receive a 10-day course of either amoxicillin or placebo. In addition, all subjects will receive an analgesic, an oral decongestant, a nasal saline spray, and an antitussive agent. Subject outcomes will be assessed by telephone interview at 0, 3, 7, 10, and 28 days. The primary outcome is the disease-specific quality of life at Day 3 measured with the SNOT-16, a validated evaluative instrument. Secondary outcomes include change in functional status and symptoms, disease recurrence, satisfaction with care and the direct costs of treatment. Tertiary outcome measures include possible subject and disease-related factors that predict clinical improvement with antibiotic treatment at Day 3 for use in future studies to aid clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be male or female, and between the ages of 18 and 70 years old.
2. The subject must have symptoms of acute bacterial rhinosinusitis.
3. The subject must be attending a participating primary care practice in the community.
4. The subject must have symptoms of acute bacterial rhinosinusitis self-assessed as moderate, severe, or very severe.
5. The subject must have access to a phone.

Exclusion Criteria:

1. The subject is less than 18 years old or more than 70 years old.
2. The subject has very mild or mild symptom severity assessed by self report.
3. The subject has an allergy to penicillin or amoxicillin.
4. The subject has received antibiotic therapy within the past 4 weeks (including chronic treatment for acne and low dose prophylactic treatment).
5. The subject has complications of sinusitis (facial edema, cellulitis, or orbital, meningeal or cerebral signs).
6. The subject is thought to require intravenous antibiotics or hospital admission.
7. The subject is pregnant. (This will be assessed by self-report. A pregnancy test will not be required).
8. The subject has a comorbidity that may impair their immune response (such as immunodeficiency disease, uncontrolled cancer, or chemotherapy or radiation treatment).
9. The subject has cystic fibrosis.
10. The subject has Type I diabetes or is taking insulin to treat diabetes.
11. The subject had prior sinus surgery.
12. The subject requires an antibiotic for a concurrent condition such as an ear infection.
13. The subject is not able to complete the study protocol because of language barriers, lack of telephone access, or other issues.
14. Any other condition that the provider feels may interfere with the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2006-10; Primary Completion 2009-05 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Garbutt, MB, ChB, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

REFERENCES:
- [Derived] Garbutt JM, Banister C, Spitznagel E, Piccirillo JF. Amoxicillin for acute rhinosinusitis: a randomized controlled trial. JAMA. 2012 Feb 15;307(7):685-92. doi: 10.1001/jama.2012.138. PMID 22337680
- [Derived] Garbutt J, Spitznagel E, Piccirillo J. Use of the modified SNOT-16 in primary care patients with clinically diagnosed acute rhinosinusitis. Arch Otolaryngol Head Neck Surg. 2011 Aug;137(8):792-7. doi: 10.1001/archoto.2011.120. PMID 21844413

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Arm: Amoxicillin 500mg tid for 10 days in addition to symptomatic treatments
Period: Overall Study
Arm/Group | Intervention Arm | Symptomatic Treatments Only
Started | 85 | 81
Day -3 Assessment | 81 | 74
Day 7 Assessment | 80 | 75
Day 10 Assessment | 81 | 71
Day 28 Assessment | 82 | 77
Completed | 81 (The number varied by day of follow-up from 80 to 82 in the intervention group.) | 74 (The number varied by day of follow-up from 71 to 77 in the symptomatic treatment only group.)
Not Completed | 4 | 7
Not completed — Unable to contact for telephone intervie | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Symptomatic Treatments Only | Total
Number analyzed (Participants) | 85 | 81 | 166
Age Continuous [Median (Full Range); unit: years] | 32 [18 to 69] | 31 [18 to 66] | 32 [18 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 52 | 106
  Male | 31 | 29 | 60

OUTCOME MEASURES:

1. Primary Outcome: SNOT-16 Score (Sino-Nasal Outcomes Test) at Day 3
Description: The Sino-Nasal Outcomes Test (SNOT-16) assesses disease-specific quality of life for acute and chronic rhinosinusitis. This brief instrument assesses 16 sinus-related symptoms and was administered by phone. The respondent reported how much they were bothered by each item considering both its severity and frequency. Response options include no problem (0), mild or slight problem (1), moderate problem (2), severe problem (3). The SNOT-16 score is the mean score from all 16 items and ranges from 0 (minimal impact) to 3 (significant impact).
Time Frame: 4 days
Population: We analysed all participants for whom we had data at Day 3. We were unable to complete the telephone interview with 11 subjects.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intervention Arm | Symptomatic Treatments Only
Number analyzed (Participants) | 81 | 74
Units on a scale | 1.12 (0.54) | 1.14 (0.55)
Statistical Analysis 1: Comparison: Intervention Arm vs Symptomatic Treatments Only; We used analysis of variance, controlling for disease severity at baseline to test the null hypothesis that there was no difference between study groups at this point in time; Test type: Superiority or Other; p = 0.83, ANOVA — The a priori threshold for statistical significnace was p less than or equal to 0.05; Adjusted for disease severity at baseline

ADVERSE EVENTS:
Arm/Group | Intervention Arm | Symptomatic Treatments Only
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/81
Other Adverse Events (participants affected / at risk) | 39/85 | 36/81
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=85) | Symptomatic Treatments Only (N=81)
Other non-serious adverse events (General disorders) | 39 (39) | 36 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No